CLINICAL TRIAL: NCT06020482
Title: Molecular Markes of Fibrosis of Single Types of Endometriosis and Their Use in Predicting Disease Severity
Brief Title: Molecular Markes of Fibrosis of Endometriosis and Their Use in Predicting Disease Severity
Acronym: MMF
Status: Recruiting | Type: Observational
Sponsor: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Zdenka Lisa, M.D., General University Hospital, Prague
Other Study IDs: GIP-23-L-03-223
Record Dates: First submitted 2023-08-28; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Molecular Markers of Fibrosis of Single Types of Endometriosis and Their Use in Predicting Disease Severity
Keywords: endometriosis, moleculars markers of fibrosis, deep infiltrating endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — specimen of eutopic endometrium and non-eutopic endometrial-like tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- A-OE: women with ovarian endometriosis (study group)
  Interventions: Other: Molecular markes of fibrosis of single types of endometriosis and their use in predicting disease severity
- A-PE: women with peitoneal endometriosis (study group)
  Interventions: Other: Molecular markes of fibrosis of single types of endometriosis and their use in predicting disease severity
- A-DE: women with deep infiltrating endometriosis (study group)
  Interventions: Other: Molecular markes of fibrosis of single types of endometriosis and their use in predicting disease severity
- B: women without endometriosis

INTERVENTIONS:
Other: Molecular markes of fibrosis of single types of endometriosis and their use in predicting disease severity — The aim of the study is to analyze molecular markers of fibrosis in female patients with endometriosis vs. without endometriosis. These features will be compared for their clinical status and progression of the disease before and after treatment. Identification and validation of these features appears to be a crucial step in predicting progression of the disease. Moreover, we would be able to modify follow-up and treatment management in high-risk patients for endometriosis.
  Groups: A-DE; A-OE; A-PE

SUMMARY:
The primary aim of the project is to analyse gene expression in individual types of ectopic endometrium (ovarian endometriosis, peritoneal endometriosis, deep infiltrating endometriosis) and compare it with gene expression in eutopic endometrium. The analysis focuses on the identification of genes with significantly increased expression in each type of ectopic endometrium and comparison of their expression with the degree of disease, ovarian reserve and clinical manifestations of the disease (pain, infertility).

DETAILED DESCRIPTION:
Endometriosis is defined as the presence of endometrial-like tissue outside the uterine cavity. It is a chronic benign estrogen-dependent disease affecting approximately 10% of women of reproductive age. It significantly affects the quality of life of affected women despite available treatment. The disease is most manifested by symptoms of pain (chronic pelvic pain, dysmenorrhea, dyspareunia, dyschesia) and sterility. In addition to adenomyosis (internal endometriosis), there are three main types of the disease - ovarian endometriosis (OE), peritoneal endometriosis (PE) and deep infiltrating endometriosis (DE). Although it is a benign disease, it shares certain characteristics with malignant diseases, such as the ability to relapse and grow infiltratively. Endometriosis tends to recur and develop adhesions and fibrotic scarring in the abdominal cavity, which means a higher risk of more severe symptoms and organ damage.

The origin of the disease remains unclear. Although it is believed that ectopic endometrial cells exhibit molecular abnormalities that promote their ability to adhere and growth outside the uterine cavity. Previous studies have identified various proteins that are up-regulated in endometrial-like tissue compared to normal endometrium, such as ACTA2, ALDH1B, FABP4 or MMP9. However, the diagnostic utility of these biomarkers is limited. In addition, there is no established biomarker that is specific to different types of ectopic endometrium or correlates with disease severity. Therefore, the identification and validation of these molecular abnormalities and proteins appears to be a key point in the effort to elucidate the pathway of disease development. This might open new possibilities for predicting disease progression so that monitoring a treatment of the disease might be tailored to the high-risk patients.

The aim of our study is to analyze molecular markers of fibrosis in eutopic and ectopic endometrium in women with endometriosis and compare them with endometrium of women without endometriosis. These markers will be correlated with the clinical state and course of disease before and after treatment. By this analysis we would like to find parameters that may correlate with the severity of the disease, risk of recurrence or postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* women (18-45 years)
* signed informed consent with the study
* absence of hormonal treatment 3 months before the planned procedure

Inclusion criteria for group A:

- laparoscopically and histologically confirmed endometriosis dg.

Inclusion criteria for group B:

* patients without endometriosis
* patients who are undergoing an elective laparoscopic or hysteroscopic procedure in our department for another benign indication
* patients with excluded malignant disease

Exclusion Criteria:

* absence of informed consent
* patients who do not meet the inclusion criteria during surgery
* patient younger than 18 years of age or older than 45 years of age

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women (18-45 years) with or without endmetriosis
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Molecular markers of fibrosis of single types of endometriosis and their use in predicting disease severity | The project is supposed to be lasting 3 years.
  The aim of our study is to analyze molecular markers of fibrosis in eutopic and ectopic endometrium in women with endometriosis and compare them with endometrium of women without endometriosis. These markers will be correlated with the clinical state and course of disease before and after treatment. By this analysis we would like to find parameters that may correlate with the severity of the disease, risk of recurrence or postoperative complications.

CONTACTS AND LOCATIONS:
Locations (1):
- General University Hospital in Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No